CLINICAL TRIAL: NCT06517043
Title: Upregulating Spinal Circuits to Enhance Balance and Walking and to Increase Spinal Excitability in Older Adults
Brief Title: Spinal Networks of Balance Learning and Retention in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202400382; R21AG084944 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Aging
Keywords: aging; balance; walking; spinal cord; electrical stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tsDCS treatment (Active Comparator): Participants will receive 30 minutes of continuous 2.5-mA tsDCS over the lumbar regions while engaging in a 30-minute complex balance task during each intervention session over a period of 2 weeks (every other day), totaling 5 intervention visits.
  Interventions: Behavioral: Balance Training; Device: Spinal Active tsDCS
- Sham tsDCS control (Sham Comparator): Participants will receive 3 minutes of 2.5-mA tsDCS over the lumbar regions while engaging in a 30-minute complex balance task during each intervention session over a period of 2 weeks (every other day), totaling 5 intervention visits.
  Interventions: Behavioral: Balance Training; Device: Spinal Sham tsDCS

INTERVENTIONS:
Behavioral: Balance Training — Complex balance task involving static and dynamic weight shifting and coordinated stepping
Device: Spinal Active tsDCS — Active tsDCS over lumbar regions
  Arms: Active tsDCS treatment
Device: Spinal Sham tsDCS — Sham tsDCS over lumbar regions
  Arms: Sham tsDCS control

SUMMARY:
Age-related balance and walking issues increase fall risks, leading to injuries, higher healthcare costs, reduced quality of life, and increased morbidity/mortality rates. Preserving functional ability is a crucial public health priority, with the potential to reduce healthcare costs and enhance older adults' quality of life. Declines in balance and walking ability threaten independence. These declines are attributed to spinal network impairments and may be mitigated by targeted interventions aimed at addressing age-related spinal cord impairment to enhance functional outcomes. However, there is a lack of research into how the aging spinal cord affects balance/walking. In older adults, the spinal cord is less excitable, conducts signals more slowly, and is subject to neural noise. Intervening on age-related impairment of the spinal cord to improve balance/walking ability is a very promising but untapped area of research. A therapeutic approach that combines dynamic balance training with non-invasive electrical spinal stimulation may be effective in preserving functional abilities. This study tests whether electrical stimulation of the spinal lumbar regions is more beneficial than sham stimulation.

DETAILED DESCRIPTION:
A high proportion of older adults are currently or soon will be at risk for the well-known decline in walking and balance abilities that occur with aging. Preserving those abilities has become a major public health priority. Balance training can enhance functional abilities or attenuate functional decline; however, age-related motor deficits may impair practice-based motor learning and behavioral performance. Due to the crucial roles of the spinal cord in balance and walking performance, it is important to consider that age-related neural impairment of the spinal cord is a likely contributing factor. Specifically, the spinal cord in older adults has fewer neurons, is less excitable, and conducts signals more slowly.

Despite ample evidence of impaired spinal cord neuronal structure and function with aging, the potential benefit of an intervention targeting spinal control of balance and walking control has been largely unexplored. This dearth of research may be due in part to the lack of a clinically feasible intervention. However, the recent emergence of transcutaneous spinal direct current stimulation (tsDCS) as a non-invasive intervention creates new opportunities for understanding spinal cord contributions to balance and walking performance. Notably, our previous study was the first demonstration of the safety and feasibility of a lab-based intervention that combined tsDCS with complex walking practice. These initial findings support the enhanced efficacy of locomotor learning during a single session when combined with tsDCS in older adults. Building on the success of this preliminary data, the investigators now propose an extended, multisession intervention that combines tsDCS with balance training. The proposed study will be among the first multi-session trial to investigate the effects of tsDCS as an adjunct therapy to dynamic balance training in older adults.

This study aims to enroll 30 older adults aged 65 years or older with balance or walking deficits, determined through objective assessments. All participants will undergo the same five-session balance training over a 2-week period, which will emphasize the use of a unique balance exergaming device called the Dividat Senso. Participants will be randomly assigned to a tsDCS adjuvant group. The "Active group" will receive 30 continuous minutes of 2.5-mA tsDCS over lumbar regions T11/T12. The "Sham group" will receive the sham protocol, which involves an identical montage and stimulation arrangement but delivers no current for 27 minutes. Each 30-minutes session will be preceded and followed by balance and walking assessments to examine the intervention's effects over time. Spinal excitability, measured via soleus H-reflex testing, will be assessed immediately before and after tsDCS at the first and last intervention. Behavioral assessments will occur at baseline, 1 day post-intervention, and 10-day post-intervention to investigate pre vs. post effects and retention intervention effects. Prefrontal activity will be measured using functional near-infrared spectroscopy (fNIRS) during the behavioral assessments to evaluate demand on executive control networks.

The objective of using tsDCS is to upregulate spinal circuits to make them more responsive to task-specific activation, thereby fostering more robust learning and consolidation to enhance performance in dynamic balance tasks. Thus, the overarching hypothesis of the proposed research is that tsDCS will be a potent adjuvant therapy to a dynamic balance intervention by reinforcing task-appropriate spinal excitation to promote skill acquisition and retention, thereby improving balance and walking. This study will focus on achieving the following specific aims:

Specific Aim 1: Acquire preliminary effect size and response variance data to assess whether active adjuvant tsDCS therapy combined with dynamic balance training enhances practice-related gains in balance and walking performance and retention over time.

Specific Aim 2: Establish evidence of increased spinal excitability following tsDCS, positively correlating with gains in balance and walking functions.

The long term deliverable of this line of research will be a clinically feasible multi-modal intervention to assist in preserving motor function and independence in older adults. The knowledge and experience gained from this study will enable us to conduct larger studies to better understand the effects of aging on the spinal cord and to test rehabilitation interventions to promote healthy aging among older adults.

ELIGIBILITY:
Inclusion Criteria:

* age range: 65 to 95 years
* no severe high blood pressure: Resting systolic < 180 mmHg and diastolic < 100 mmHg
* no severe vision impairment: Visual acuity ≥ 20/70 as determined by Snellen eye chart
* walking problem: Preferred walking speed slower than 1.0 m/s over 10 meters
* balance problem: Berg Balance Scale score < 45
* no cognitive impairment: Montreal Cognitive Assessment (MoCA) score ≥ 26 out of 30

Exclusion Criteria:

* diagnosed neurological disorder or injury of the central nervous system, or observation of symptoms consistent with such a condition (Alzheimer's, Parkinson's, stroke, etc.)
* severe arthritis, such as awaiting joint replacement
* current cardiovascular, lung or renal disease; untreated diabetes; terminal illness
* myocardial infarction or major heart surgery in the previous year
* cancer treatment in the past year, except for nonmelanoma skin cancers and cancers having an excellent prognosis (e.g., early stage breast or prostate cancer)
* current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* currently taking medications that affect the central nervous system, such as benzodiazepines, anti-cholinergic medication, and GABAergic medication, among others
* uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* bone fracture or joint replacement in the previous six months
* current enrollment in any other clinical trial
* planning to relocate out of the area during the study period
* non-English* speaking, due to the likelihood of difficulties following instructions and communicating remotely
* clinical judgment of the investigative team

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Center of Pressure (COP) balance control | Baseline, 1-day post-intervention (after intervention), 10-day follow-up (after post-intervention)
  Change in the center of pressure during static and dynamic postural control on a Dividat Senso pressure-sensitive plate will be assessed from baseline to post-intervention and follow-up.
Walking speed over obstacle course | Baseline, 1-day post-intervention (after intervention), 10-day follow-up (after post-intervention)
  Change in fastest walking speed over a 10-meter obstacle course on the GAITRite system will be assessed from baseline to post-intervention and follow-up.
Spinal excitability via Soleus H-reflex testing | Baseline and immediately following 30-minute intervention
  Change in spinal excitability, measured via the soleus H-reflex testing using electromyography, will be assessed before and immediately following active or sham tsDCS (combined with balance training) during the 1st and 5th of the total five intervention sessions. The magnitude of change will be compared between these sessions.

SECONDARY OUTCOMES:
Score on standardized balance assessment (Berg Balance Scale) | Baseline, 1-day post-intervention (after intervention), 10-day follow-up (after post-intervention)
  Change in balance scores will be assessed using the Berg Balance Scale from baseline to post-intervention and follow-up. The scale ranges from 0 to 56, with higher scores indicating better balance performance.
Score on standardized walking assessment (Functional Gait Assessment) | Baseline, 1-day post-intervention (after intervention), 10-day follow-up (after post-intervention)
  Change in walking scores will be assessed using the Functional Gait Assessment from baseline to post-intervention and follow-up. The scale ranges from 0 to 30, with higher scores indicating better walking performance.
Completion time on test of executive function (Trail Making Test) | Baseline, 1-day post-intervention (after intervention), 10-day follow-up (after post-intervention)
  Change in completion time from baseline to post-intervention and follow-up will be assessed using the Trail Making Test. Shorter times indicate better cognitive performance.
tsDCS treatment-related adverse events as assessed by a survey questionnaire. | Baseline and following 30-minute intervention
  Change in the score of side effects from tsDCS (e.g., sensations of burning, tingling, itching, and pain) will be assessed before and following active or sham tsDCS (combined with balance training) for every 30-minute intervention session using a survey questionnaire. Each question on the scale ranges from 0 to 10, and the scores will be averaged. A higher mean score indicates a higher severity of side effects.
Prefrontal cortical activity using fNIRS | Baseline, 1-day post-intervention (after intervention), 10-day follow-up (after post-intervention)
  Change in prefrontal brain activity during static and dynamic balance control and fastest walking assessments will be assessed using functional Near-Infrared Spectroscopy (fNIRS) from baseline to post-intervention and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Malcom Randall VA Medical Center Brain Rehabilitation Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset will be created and shared pursuant to a Data Use Agreement appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
Supporting Information: Study Protocol, CSR
Time Frame: The Limited Dataset will be completed after the study is completed and primary/secondary data accepted for publication.